CLINICAL TRIAL: NCT00969046
Title: EPO906 Phase I 6-arm Trial to Optimize Administration Exploring Single Dose Bolus and Continuous Infusion Over 1 or 5 Days Every 3 or 4 Weeks in Patients With Pretreated Advanced Colon Cancer With Nutritional Support Treatment and Intensive Management of Diarrhea
Brief Title: Dose-Escalation Study in Advanced Colon Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEPO906A2117
Record Dates: First submitted 2009-08-10; First posted 2009-08-31 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2016-04

CONDITIONS: Colon Cancer
Keywords: Colon cancer; MTD; DLT; EPO906; patupilone
MeSH Terms: conditions — Colonic Neoplasms | interventions — epothilone B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bolus (Experimental): 20 min bolus infusion
  Interventions: Drug: EPO906 (patupilone)
- CIV-1d (Experimental): 1 day continuous infusion
  Interventions: Drug: EPO906 (patupilone)
- CIV-5d (Experimental): 5 day continuous infusion
  Interventions: Drug: EPO906 (patupilone)

INTERVENTIONS:
Drug: EPO906 (patupilone)

SUMMARY:
This study is exploring different administration schedules (short versus prolonged infusion) to optimize the safety and efficacy profile of EPO906A (patupilone) in patients with pretreated advanced colon cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, locally advanced, progressive or metastatic colon cancer, up to 4 prior lines of prior chemotherapy, at least one measurable lesion according to RECIST
2. Age ≥ 18 years
3. Life expectancy ≥ 12 weeks
4. WHO performance status of 0-1
5. Negative serum pregnancy test
6. Adequate hepatic or renal function and hematological parameters

Exclusion Criteria:

1. Brain metastases
2. Ileostomy or colonostomy
3. History of pelvic radiotherapy
4. Grade > 1 diarrhea at baseline

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-11; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To identifymaximum tolerated dose (MTD) | During cycle 1 and 2 (approx 6 to 8 wks)

SECONDARY OUTCOMES:
To characterize the safety and tolerability of patupilone by assessing adverse events (AEs) and serious adverse events (SAEs), hematology and biochemistry labs, vital signs, performance status, and by physical/neurological exams | at base line, every 3 weeks prior to start of the next dose, at end of treatment
To evaluate preliminary anti-tumor activity of patupilone using standard imaging technologies (e.g. best overall response rate and time to progression according to Response Evaluation Criteria in Solid Tumors [RECIST]) | at baseline and every 8 wks
To evaluate the blood concentrations profile (pharmacokinetics [PK]) of patupilone by multiple blood sampling before, during and after drug administration | Cycle 1 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Royal London Hospital
Locations (6):
- Czechia (2):
  - Novartis Investigative Site, Hradec Králové
  - Novartis Investigative Site, Prague
- France (2):
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Toulouse
- Novartis Investigative Site, Barcelona, Spain
- Novartis Investigative Site, London, United Kingdom

REFERENCES:
- See also: Results for CEPO906A2117 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2945